CLINICAL TRIAL: NCT03581539
Title: Randomized, Prospective, Study Comparing Four-quadrant Transverses Abdominis Plane (TAP) Block, Quadratus Lumborum (QL) Block and Surgeon Infiltration Using Exparel for Postoperative Analgesia After Laparoscopic Nephrectomy
Brief Title: Comparing 3 Different Types of Pain Blocks After Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kevin Michael Backfish-White, Anesthesiologist, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1801979369
Record Dates: First submitted 2018-06-13; First posted 2018-07-10 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Nephrectomy
Keywords: Laparoscopic Nephrectomy,; Simple Nephrectomy; Partial Nephrectomy; Pain,acute; Pain,postoperative
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Patients randomized to four-quadrant Transverses Abdominis Plane (TAP) block, Quadratus Lumborum (QL) block or surgeon infiltration using Exparel for postoperative analgesia after laparoscopic nephrectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group #1 (Active Comparator): Transverses Abdominis Plane (TAP) block
  Interventions: Procedure: Transverses Abdominis Plane (TAP) block
- Group #2 (Active Comparator): Quadratus Lumborum (QL) block
  Interventions: Procedure: Quadratus Lumborum (QL) block
- Group #3 (Active Comparator): Surgeon Infiltration using Exparel
  Interventions: Procedure: Surgeon Infiltration using Exparel

INTERVENTIONS:
Procedure: Transverses Abdominis Plane (TAP) block — TAP block - Participants will get an injection of bupivacaine and exparel (numbing medicine) in the four different locations of your stomach. To be more specific, the injection placed between your oblique muscles in four different locations right after you are asleep and just before the start of surgery. Investigators will use an ultrasound machine (the machine works by taking pictures of internal organs by bouncing sound waves off them and recording the echoes) to find the abdominal muscle layers and find the correct location to inject the numbing medicine between the muscle layers.
  Arms: Group #1
Procedure: Quadratus Lumborum (QL) block — QL block - Participants will get an injection of bupivacaine with exparel (numbing medicine) in two locations in your lower stomach. To be more specific, an injection will take place inside your quadratus lumborum muscle which is slightly deeper than your oblique muscles right after you are asleep and right before surgery. Investigators will use an ultrasound machine (the machine works by taking pictures of internal organs by bouncing sound waves off them and recording the echoes) to find the abdominal muscle layers and find the correct location to inject the numbing medicine between the muscle layers.
  Arms: Group #2
Procedure: Surgeon Infiltration using Exparel — SI group - at the end of the surgery and just prior to you waking up, the surgeon will use a needle to inject the surgical incision site with bupivacaine and exparel (numbing medicine) spreading the medicine evenly as the needle is slowly withdrawn to make sure all layers are evenly filled with the medicine that will numb the area.
  Arms: Group #3

SUMMARY:
All three methods of postoperative analgesia have been shown to decrease postoperative pain control in nephrectomy patients, the three methods have never been compared to each other.

This study aims to compare three different pain techniques proven to be beneficial in surgical nephrectomies, including the efficacy and the side effects of each technique.

DETAILED DESCRIPTION:
Both four-quadrant TAP block and QL blocks will be done after induction of anesthesia but prior to incision. Surgeon infiltration will be completed intraoperatively at the end of the surgery. All procedures will be done using sterile technique with masks, hats, and sterile gloves. All procedures will be placed under the supervision of the attending anesthesiologist on the acute pain service.

All patients will receive 1 gm acetaminophen and 600 mg gabapentin preoperatively per SOC. Patients above 70 years will receive 300 mg gabapentin per SOC. Patients will be grouped by type of nephrectomy: simple, radical, or partial. Patients will be randomized to type of block. Intraoperatively, the patient will receive ketamine 0.5 mg/kg LBM at the beginning of the case followed by a 0.25 mg/kg/hr infusion during surgery but turned off prior to emergence per SOC; patients with relative contraindications to ketamine such as history of seizures may not receive ketamine and this will NOT be considered a deviation.

For group 1, the TAP block group, after the patient is induced, the skin will be prepped with ChloPrep and a clean, sterile transducer will be placed in an axial (transverse) plane to visualize the TAP plane just superior to the iliac crest. This will allow us to identify the three muscular layers of the abdominal wall: the external oblique (most superficial), the internal oblique, and the transversus abdominis. Using an in-plane technique (seeing the needle at all times), the needle will be advanced into the fascial plane between the internal oblique and transversus abdominis muscles under ultrasound guidance and 15 mL 0.125% bupivacaine plus 5 mL of Exparel® will be injected into the fascial plane; this procedure will be repeated in the other four quadrants of the abdomen. The tip of the needle will be observed under ultrasound at all times, making this a minimal risk procedure. It is also important to note that the mg dose of bupivacaine with exparel will never be in a ratio greater than 1:2 per Exparel dosing guidelines. A total of 80 mL will be given.

The QL block will be performed after induction with the patient placed in a slight lateral position in order to facilitate visualization of the Quadratus Lumborum muscle. Once the skin has been prepped and the sterile transducer is applied, the continuation of the transversalis fascia will be visualized along with the termination of the external and internal obliques. The quadratus lumborum will be identified deep to these structures. Once identified, an in plane technique will be used in order to place the needle in the plane just superior to the QL and 20 mL of 0.125% bupivacaine along with 10mL of Exparel will be injected. The same process will be repeated on the contralateral side. Once again the needle will be visualized throughout the procedure.

Surgeon infiltration will be completed at the end of the procedure before the patient emerges from general anesthesia. The needle will be inserted approximately 0.5 to 1 cm into the tissue plane to ensure that all layers of the surgical incision are infiltrated. The local anesthetic solution of 5 mL 0.125% bupivacaine plus 10 mL Exparel® will be injected while slowly withdrawing the needle to decrease the risk of intravascular injection.22 A total of 30 mL will be delivered. Surgeon name will be recorded.

All patients will be scheduled on PO acetaminophen and PO gabapentin daily postoperatively per SOC. PO oxycodone or tramadol PRN per SOC will be started once patients are tolerating a diet. PRN IV dilaudid, fentanyl, or morphine will also be given for severe breakthrough pain per SOC.

Opioid usage at 1, 24, 48 and 72 hours after the block will be recorded by a member of the research team. Pain scores at rest and on movement will be measured using Visual Analog Scale (VAS). Nausea will be measured using a categorical scoring system (none=0; mild=1; moderate=2; severe=3). Sedation scores will also be assessed by a member of the study team using a sedation scale (awake and alert=0; quietly awake=1; asleep but easily roused=2; deep sleep=3). All these parameters will be measured at 1, 24, 48 and 72 hours after the epidural or PVB. Investigators will record postoperative time of 1st flatus. Patients will be encouraged to ambulate on postoperative day 1 under supervision. Their ambulation activity will be recorded. First liquid and first food intake will also be recorded.

All patients will receive a phone call approximately two weeks after surgery for assessment for patient satisfaction and pain scores. Patients will be assessed by a member of the research team over the phone. They will be assessed on their pain score, opiate usage, and activity of daily living. Study participation will conclude after the two week follow-up and the questionnaire has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic nephrectomy including partial, simple and radical nephrectomy
* ASA class 1, 2, 3 or 4
* Age 18 or older, male or female

Exclusion Criteria:

* Any contraindication for TAP block, QL block or surgeon infiltration
* Donor Nephrectomy
* History of substance abuse in the past 6 months
* Patients on more than 30mg po morphine equivalents of opioids, staff anesthesiologist will confirm this portion prior to enrollment.
* Any physical, mental or medical conditions which in the opinion of the investigators, may confound quantifying postoperative pain resulting from surgery.
* Known allergy to bupivacaine or Exparel
* Patients <40kg or >110 kg TBW

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Primary endpoint of this study will be VAS pain score at 24 hours | Pain scores will be measured 24 hours after surgery
  The VAS scores will be taken with both rest and movement (knee flexion) and will be measured by a study team investigator using Visual Analog Scale (VAS). Using a scale of 1-10 for documentation with 10 being the worst pain and 0 being no pain
Primary endpoint of this study will be VAS pain score at 48 hours | Pain scores will be measured 48 hours after surgery
  Pain scores will be measured by a study team investigator using Visual Analog Scale (VAS). Using a scale of 1-10 for documentation with 10 being the worst pain and 0 being no pain

SECONDARY OUTCOMES:
Secondary endpoint includes total IV and PO (By Mouth) opioid consumption at 72 hours | Opioid consumption will be measured at 1 hour post op, 24, 48, and 72 hours post op. The total amount will be recorded
  Opioid consumption will be collected by a study team member post-operatively up to 3 days per protocol time requirements

OTHER OUTCOMES:
Average Nausea scores over 72 hours | Nausea scores will be documented at 1 hour post op, 24, 48, and 72 hours after the block. The scores will then be averaged
  Nausea scores will be collected by a study team member post operatively up to 3 days per protocol. Nausea will be recorded as none, mild, moderate or severe
Average Sedation scores over 72 hours | Sedation scores will be documented at 1 hour post op, 24, 48, and 72 hours after the block. The scores will then be averaged
  Sedation scores will be documented by a study team member post operatively up to 3 days per protocol requirements. Determining if patient is awake and alert, quietly awake, asleep and arousable, or deep sleep
Subjects overall satisfaction scores | Post operatively at hour 24
  Subjects will be followed up to 24 hours post operatively by a study team member to document patient overall satisfaction scores
Subjects overall satisfaction scores | Post operatively at hour 48
  Subjects will be followed up to 48 hours post operatively by a study team member

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Backfish-White, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States